CLINICAL TRIAL: NCT00915733
Title: Comparison of Platelet Inhibitory Effect With Adjunctive Cilostazol Versus High Maintenance-dose ClopidogrEL in Acute Myocardial Infarction Patients According to CYP2C19 Polymorphism
Brief Title: Adjunctive Cilostazol Versus High Maintenance-dose ClopidogrEL in Acute Myocardial Infarction (AMI) Patients According to CYP2C19 Polymorphism
Acronym: ACCELAMI2C19
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gyeongsang National University Hospital (Other)
Responsible Party: In-Suk Kim, Assistant Professor, Gyeongsang National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACCEL-AMI-2C19
Record Dates: First submitted 2009-06-05; First posted 2009-06-08 (Estimated); Last update posted 2009-11-10 (Estimated); Status verified 2009-11

CONDITIONS: Myocardial Infarction
Keywords: acute myocardial infarction; inhibition of platelet aggregation; triple antiplatelet therapy; high maintenance-dose clopidogrel.; CYP2C19 polymorphism; High posttreatment platelet reactivity; Platelet Aggregation Inhibitors; CYP2C19, human
MeSH Terms: conditions — Myocardial Infarction | interventions — Cilostazol; Clopidogrel; Cytochrome P-450 CYP2C19; CYP2C19 protein, human; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- triple group (Active Comparator): Additive cilostazol to dual antiplatelet therapy (triple antiplatelet therapy) in patients with acute myocardial infarction (AMI).
  Received cilostazol 100 mg twice daily in addition to aspirin 100 mg and clopidogrel 75 mg once daily.
  Interventions: Drug: cilostazol; Drug: clopidogrel (Plavix); Genetic: CYP2C19; Drug: aspirin (Acetylsalicylic acid)
- high maintenance dose group (Active Comparator): High maintenance dose dual antiplatelet therapy in patients with acute myocardial infarction (AMI).
  Received clopidogrel 150 mg/day with aspirin 100 mg once daily.
  Interventions: Drug: clopidogrel (Plavix); Genetic: CYP2C19; Drug: aspirin (Acetylsalicylic acid)

INTERVENTIONS:
Drug: cilostazol — 100 mg twice daily for at least 1 month
  Other Names: Otsuka brand of cilostazol
  Arms: triple group
Drug: clopidogrel (Plavix) — 150 mg once daily (high maintenance dose group arm), 75 mg once daily (triple group arm)
  Other Names: Plavix
Genetic: CYP2C19 — CYP2C19 polymorphism study: Two CYP2C19 polymorphisms, CYP2C19*2 (rs4244285, c. 681G>A, p.P227P), and CYP2C19*3 (rs4986893, c. 636G>A, p. W212X), are investigated using the ABI SNaPshot reaction and the ABI 3100 automated genetic analyzer.
  Other Names: Cytochrome 2C19
Drug: aspirin (Acetylsalicylic acid) — aspirin 100 mg qd
  Other Names: Acetylsalicylic acid

SUMMARY:
Percutaneous coronary intervention (PCI) with stent implantation is the preferred reperfusion strategy for treatment of acute myocardial infarction (AMI). Despite advances in both devices and pharmacological support for AMI patients undergoing PCI, the risk of recurrent ischemic events has been higher than that of elective PCI. Among therapeutic options for surmounting clopidogrel hyporesponsiveness, higher loading doses and maintenance doses of clopidogrel achieved significant enhancements in the speed of onset and intensity of inhibition and these approaches have been widely adapted in clinical practice. Interestingly, recent studies found that carriers of the loss-of-function hepatic cytochrome (CYP) 2C19 allele had significantly lower levels of the active metabolite of clopidogrel, diminished platelet inhibition, and a higher rate of major adverse cardiovascular events than did non-carriers, in the setting of PCI and acute coronary syndrome (ACS). These findings raise the need of solutions to overcome enhanced post-clopidogrel platelet reactivity by the influence of the loss-of-function CYP2C19 allele. Increasing the dose of clopidogrel, new potent P2Y12 antagonists (such as prasugrel), or other antiplatelet drugs such as cilostazol may be alternative antiplatelet regimens in patients with the loss-of-function CYP variant. A recent study demonstrated that adjunctive cilostazol to dual antiplatelet therapy (triple antiplatelet therapy) intensified platelet inhibition as compared with a high maintenance-dose (MD) of 150 mg/day. Therefore, triple antiplatelet therapy could also be an alternative antiplatelet therapy to improve platelet inhibition and clinical outcomes in carriers of CYP2C19 mutant allele.

The purpose of this study was to determine the impact of adjunctive cilostazol on platelet inhibition in carriers and non-carriers of the loss-of-function CYP2C19 allele. The investigators compared the enhanced inhibition of platelet aggregation by adjunctive cilostazol 100 mg twice daily versus high-MD clopidogrel 150 mg/day in AMI patients treated with emergent coronary stenting, according to the CYP2C19 polymorphism.

DETAILED DESCRIPTION:
* Study timeline: Enrollment period - 6 months (2009. 5.- 2009. 10.) (Follow-up period - 1 month after randomization)

  * Stenting, adjunct drug therapy and markers of myonecrosis

    1) PCI

    (1) All interventions are performed according to current standard guidelines. (2) Aspiration thrombectomy is dependent on the operator's discretion. (3) If the patients have multiple lesions, culprit lesion coverage is recommended if possible.

    (4) Any kind of DES is permitted for PCI. If the bare-metal stent is needed, it is permitted.

    (5) Direct stenting or predilation is left to the operator's decision.

    2) Antithrombotic medications
    1. Anticoagulation is begun before PCI and performed with low-molecular-weight heparin (enoxaparin) or unfractionated heparin at physician's discretion.
    2. Only tirofiban is administered if and glycoprotein IIb/IIIa inhibitors (GPI) are needed.

    3) Markers of myonecrosis

    (1) Blood samples are routinely obtained from all patients before and after PCI for assessment of CK-MB at 8, 24, 48 and 72 hours.

    (2) In case of elevated values, measurements are repeated every 12 hours until a peak value reaches or values are normalized.
    * Assays of platelet function 1) Blood sampling.

      1. Peripheral venous blood samples are drawn from an antecubital vein using a 21-gauge needle.
      2. Blood samples are collected using the double-syringe technique, in which the first 2 to 4 ml of blood is discarded to avoid spontaneous platelet activation.

      2) Light transmittance aggregometry (LTA)
      1. Blood samples are drawn into Vacutainer tubes containing 0.5 mL of sodium citrate 3.2% (Becton-Dickinson, San Jose, CA, USA) and processed within 60 minutes.
      2. Platelet-rich plasma (PRP) was obtained as a supernatant fluid after centrifuging blood at 800 rpm for 10 min. The remaining blood was further centrifuged at 2,500 rpm for 10 min to prepare platelet-poor plasma (PPP). PRP is adjusted to platelet counts of 250,000/μL by adding PPP as needed.
      3. Platelet aggregation is assessed at 37℃ using a PACKS-4 aggregometer (Helena Laboratories Corp., Beaumont, Texas, USA). Light transmission is adjusted to 0% with PRP and to 100% PPP for each measurement.
      4. Platelet aggregation is systematically measured after the addition of ADP at concentrations of 5 and 20 μM. Curves were recorded for 6 minutes.
      5. Aggregation is measured at by laboratory personnel blinded to group assignment.
      6. Absolute reduction of aggregation values (∆ Aggmax or Agglate) is defined as change of aggregation between pre-procedure and 30-day therapy:

         * Agg = pre-procedure Agg - Agg after 30-day therapy
      7. Inhibition of platelet aggregation (IPA) is defined as relative change in aggregation values (Aggmax and Agglate) between pre-procedure and 30-day therapy:

         IPA (%) = [(pre-procedure Agg - Agg after 30-day therapy)/pre-procedure Agg] X 100

      3) Rapid platelet function assay (RPFA: the VerifyNow P2Y12 assay)
      1. A point-of-care system (VerifyNow; Accumetrics, San Diego, California) is an automated turbidimetric whole blood assay based on the ability of activated platelets using cartridges containing fibrinogen-coated beads and platelet agonists.
      2. Blood is drawn into a Greiner Bio-One 3.2% citrate vacuette tube.
      3. The channel contains fibrinogen-coated polystyrene beads and 20 μM ADP as platelet agonist. This channel also contains 22 nmol/l PGE1 to suppress intracellular free calcium levels and thereby reduce the non-specific contribution of P2Y1 receptors.
      4. Results are reported in P2Y12 reaction units (PRU).
      5. Absolute reduction of PRU is defined as change of PRU between pre-procedure and 30-day therapy:

         ∆ PRU = pre-procedure PRU - PRU after 30-day therapy
      6. Percent inhibition (PI) of PRU is defined as relative change between pre-procedure and 30-day therapy:

         PI (%) = [(pre-procedure PRU - PRU after 30-day therapy)/pre-procedure PRU] X 100

         2-8. CYP2C19 genotyping

      <!-- -->

      1. CYP2C19 genotype is determined by a polymerase chain reaction (PCR). SNaPshot method, using genomic DNA isolated from leukocytes of peripheral venous blood with an extraction kit (QIAampR DNA Blood Mini Kit, Qiagen, Hilden,Germany).
      2. Two CYP2C19 polymorphisms, CYP2C19*2 (rs4244285, c. 681G>A, p.P227P), and CYP2C19*3 (rs4986893, c. 636G>A, p. W212X), are investigated using the ABI SNaPshot reaction and the ABI 3100 automated genetic analyzer (Applied Biosystems, Foster City, CA, USA).

         ****Statistics and Data analysis

      <!-- -->

      1. Sample Size Estimation

         @ based on previous our study(ACCEL-AMI)

         Absolute reduction of 5 μM ADP-induced maximal aggregation by adjunctive cilostazol after 30 days : 24.0%

         Absolute reduction of 5 μM ADP-induced maximal aggregation by adjunctive high dose maintenance clopidogrel 150mg/day after 30 days : 11.0%

         Relative difference of enhanced platelet inhibition between two regimens :

         54.0% - Two-sided α-level = 0.05 - Power = 95% - Triple group: high-MD group = 1: 1 - Standard deviation = 0.4

         At least 15 patients per each group were required.

         @ based on previous another study(CYP2C19 polymorphism study)

         The ratio of Korean patients carrying wild type CYP2C19 vs mutant type=4:6

         The required patients of wild type group : 15 patients The required patients of mutant type group : 23 patients

         Final required patients (15+23)*2=76 patients
      2. Analysis Continuous variables are presented as means ± SD and compared using Student unpaired t or Mann-Whitney U tests. Categorical variables are presented as numbers or percentages and were compared using chi-square or Fisher's exact tests (if an expected frequency was < 5). The characteristics and platelet function measures of the 3 groups were analyzed by Friedman's repeated ANOVA on ranks. After demonstration of significant differences among variables by ANOVA, post hoc comparisons between therapy pairs were made with the Student-Newman-Keuls procedure for multiple comparisons. A p value < 0.05 was considered to indicate a significant difference. Statistical analysis was performed using commercially available software (SPSS version 13; SPSS Inc., Chicago, Illinois, USA).
      3. Data modulation DSMB (Data Safety Monitoring Board) CEC (Clinical Event Committee)

ELIGIBILITY:
Inclusion Criteria:

1. The patient must be at least 18 years of age.
2. clinical symptoms compatible with acute myocardial ischemia within 12 h before admission with a subsequently documented increase in cardiac markers.
3. Measured pre-discharge platelet reactivity in case of normalized CK-MB value after coronary stenting.

Exclusion Criteria:

1. A history of active bleeding and bleeding diatheses.
2. Oral anticoagulation therapy with coumadin.
3. Contraindication to antiplatelet therapy.
4. LV ejection fraction < 30% or NYHA 3/4.
5. Leukocyte count < 3,000/mm3 and/or platelet count < 100,000/mm3.
6. AST or ALT ≥ 3 times upper normal.
7. Serum creatinine level ≥ 2.5 mg/dl.
8. Stroke within 3 months.
9. Non-cardiac disease with a life expectancy < 1 year.
10. Inability to follow the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2009-05; Primary Completion 2009-10 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Absolute reduction of maximal platelet aggregation (Aggmax) by 5 & 20 μM ADP induced LTA | 30 days

SECONDARY OUTCOMES:
Absolute reduction of late platelet aggregation (Agglate) by 5 & 20 μM ADP induced LTA | 30 days
Absolute reduction of P2Y12 reaction unit (PRU) | 30 days
The rate of high post-treatment platelet reactivity | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: In-Suk Kim, MD.PhD., Principal Investigator — Gyeongsang National University Hospital
Locations (1):
- Gyeongsang National University Hospital, Jinju, South Korea

REFERENCES:
- [Result] Jeong YH, Lee SW, Choi BR, Kim IS, Seo MK, Kwak CH, Hwang JY, Park SW. Randomized comparison of adjunctive cilostazol versus high maintenance dose clopidogrel in patients with high post-treatment platelet reactivity: results of the ACCEL-RESISTANCE (Adjunctive Cilostazol Versus High Maintenance Dose Clopidogrel in Patients With Clopidogrel Resistance) randomized study. J Am Coll Cardiol. 2009 Mar 31;53(13):1101-9. doi: 10.1016/j.jacc.2008.12.025. PMID 19324253
- [Result] Kim IS, Choi BR, Jeong YH, Kwak CH, Kim S. The CYP2C19*2 and CYP2C19*3 polymorphisms are associated with high post-treatment platelet reactivity in Asian patients with acute coronary syndrome. J Thromb Haemost. 2009 May;7(5):897-9. doi: 10.1111/j.1538-7836.2009.03319.x. Epub 2009 Feb 12. No abstract available. PMID 19220726
- [Result] Mega JL, Close SL, Wiviott SD, Shen L, Hockett RD, Brandt JT, Walker JR, Antman EM, Macias WL, Braunwald E, Sabatine MS. Cytochrome P450 genetic polymorphisms and the response to prasugrel: relationship to pharmacokinetic, pharmacodynamic, and clinical outcomes. Circulation. 2009 May 19;119(19):2553-60. doi: 10.1161/CIRCULATIONAHA.109.851949. Epub 2009 May 4. PMID 19414633
- [Result] Collet JP, Hulot JS, Pena A, Villard E, Esteve JB, Silvain J, Payot L, Brugier D, Cayla G, Beygui F, Bensimon G, Funck-Brentano C, Montalescot G. Cytochrome P450 2C19 polymorphism in young patients treated with clopidogrel after myocardial infarction: a cohort study. Lancet. 2009 Jan 24;373(9660):309-17. doi: 10.1016/S0140-6736(08)61845-0. Epub 2008 Dec 26. PMID 19108880
- [Result] Mega JL, Close SL, Wiviott SD, Shen L, Hockett RD, Brandt JT, Walker JR, Antman EM, Macias W, Braunwald E, Sabatine MS. Cytochrome p-450 polymorphisms and response to clopidogrel. N Engl J Med. 2009 Jan 22;360(4):354-62. doi: 10.1056/NEJMoa0809171. Epub 2008 Dec 22. PMID 19106084
- [Result] Lee SW, Park SW, Kim YH, Yun SC, Park DW, Lee CW, Hong MK, Kim HS, Ko JK, Park JH, Lee JH, Choi SW, Seong IW, Cho YH, Lee NH, Kim JH, Chun KJ, Park SJ. Drug-eluting stenting followed by cilostazol treatment reduces late restenosis in patients with diabetes mellitus the DECLARE-DIABETES Trial (A Randomized Comparison of Triple Antiplatelet Therapy with Dual Antiplatelet Therapy After Drug-Eluting Stent Implantation in Diabetic Patients). J Am Coll Cardiol. 2008 Mar 25;51(12):1181-7. doi: 10.1016/j.jacc.2007.11.049. PMID 18355656
- [Result] Lee BK, Lee SW, Park SW, Lee SW, Park DW, Kim YH, Lee CW, Hong MK, Kim JJ, Jang S, Chi HS, Park SJ. Effects of triple antiplatelet therapy (aspirin, clopidogrel, and cilostazol) on platelet aggregation and P-selectin expression in patients undergoing coronary artery stent implantation. Am J Cardiol. 2007 Aug 15;100(4):610-4. doi: 10.1016/j.amjcard.2007.03.070. Epub 2007 Jun 29. PMID 17697815
- [Result] Lee SW, Park SW, Hong MK, Kim YH, Lee BK, Song JM, Han KH, Lee CW, Kang DH, Song JK, Kim JJ, Park SJ. Triple versus dual antiplatelet therapy after coronary stenting: impact on stent thrombosis. J Am Coll Cardiol. 2005 Nov 15;46(10):1833-7. doi: 10.1016/j.jacc.2005.07.048. Epub 2005 Oct 19. PMID 16286167
- [Result] Angiolillo DJ, Capranzano P, Goto S, Aslam M, Desai B, Charlton RK, Suzuki Y, Box LC, Shoemaker SB, Zenni MM, Guzman LA, Bass TA. A randomized study assessing the impact of cilostazol on platelet function profiles in patients with diabetes mellitus and coronary artery disease on dual antiplatelet therapy: results of the OPTIMUS-2 study. Eur Heart J. 2008 Sep;29(18):2202-11. doi: 10.1093/eurheartj/ehn287. Epub 2008 Jun 21. PMID 18567918
- [Result] Angiolillo DJ, Shoemaker SB, Desai B, Yuan H, Charlton RK, Bernardo E, Zenni MM, Guzman LA, Bass TA, Costa MA. Randomized comparison of a high clopidogrel maintenance dose in patients with diabetes mellitus and coronary artery disease: results of the Optimizing Antiplatelet Therapy in Diabetes Mellitus (OPTIMUS) study. Circulation. 2007 Feb 13;115(6):708-16. doi: 10.1161/CIRCULATIONAHA.106.667741. Epub 2007 Jan 29. PMID 17261652
- [Derived] Jeong YH, Abadilla KA, Tantry US, Park Y, Koh JS, Kwak CH, Hwang JY, Gurbel PA. Influence of CYP2C19*2 and *3 loss-of-function alleles on the pharmacodynamic effects of standard- and high-dose clopidogrel in East Asians undergoing percutaneous coronary intervention: the results of the ACCEL-DOUBLE-2N3 study. J Thromb Haemost. 2013 Jun;11(6):1194-7. doi: 10.1111/jth.12200. No abstract available. PMID 23517020
- [Derived] Jeong YH, Tantry US, Park Y, Kwon TJ, Park JR, Hwang SJ, Bliden KP, Koh EH, Kwak CH, Hwang JY, Kim S, Gurbel PA. Pharmacodynamic effect of cilostazol plus standard clopidogrel versus double-dose clopidogrel in patients with type 2 diabetes undergoing percutaneous coronary intervention. Diabetes Care. 2012 Nov;35(11):2194-7. doi: 10.2337/dc11-2351. Epub 2012 Jul 26. PMID 22837373
- [Derived] Kim IS, Jeong YH, Park Y, Yoon SE, Kwon TJ, Park JR, Hwang SJ, Koh EH, Kwak CH, Hwang JY, Kim S. Interaction analysis between genetic polymorphisms and pharmacodynamic effect in patients treated with adjunctive cilostazol to dual antiplatelet therapy: results of the ACCEL-TRIPLE (Accelerated Platelet Inhibition by Triple Antiplatelet Therapy According to Gene Polymorphism) study. Br J Clin Pharmacol. 2012 Apr;73(4):629-40. doi: 10.1111/j.1365-2125.2011.04131.x. PMID 22007612
- [Derived] Kim IS, Jeong YH, Park Y, Park KS, Yun SE, Park JR, Hwang SJ, Koh EH, Kwak CH, Hwang JY, Kim S. Platelet inhibition by adjunctive cilostazol versus high maintenance-dose clopidogrel in patients with acute myocardial infarction according to cytochrome P450 2C19 genotype. JACC Cardiovasc Interv. 2011 Apr;4(4):381-91. doi: 10.1016/j.jcin.2010.12.010. PMID 21511217
- [Derived] Jeong YH, Kim IS, Park Y, Kang MK, Koh JS, Hwang SJ, Kwak CH, Hwang JY. Carriage of cytochrome 2C19 polymorphism is associated with risk of high post-treatment platelet reactivity on high maintenance-dose clopidogrel of 150 mg/day: results of the ACCEL-DOUBLE (Accelerated Platelet Inhibition by a Double Dose of Clopidogrel According to Gene Polymorphism) study. JACC Cardiovasc Interv. 2010 Jul;3(7):731-41. doi: 10.1016/j.jcin.2010.05.007. PMID 20650435